CLINICAL TRIAL: NCT01673165
Title: A Comparison of the Effectiveness of Fortified Skimmed Mother's Milk Versus Specialized Formula in the Management of Chylous Effusion in Infants Following Cardiothoracic Surgery
Brief Title: Fortified Skimmed Mother's Milk in the Management of Chylothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Cindi Farnstrom, Certified Pediatric Nurse Practitioner, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gerber7747
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2014-10

CONDITIONS: Chylous Pleural Effusion Following Cardiothoracic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specialized Formula (Active Comparator): 25 infants of mothers who do not have breast milk or do not want to use the skimming technique. These infants will receive our standard of care - specialized formula for the treatment of chylothorax
  Interventions: Other: Specialized Formula
- Skimmed mother's milk (Experimental): 25 infants of mothers who have breast milk and who also want to learn the skimming technique will be taught the technique. The infants will then receive the skimmed breast milk for the treatment of chylothorax
  Interventions: Other: Skimmed mother's milk

INTERVENTIONS:
Other: Skimmed mother's milk — Fortified skimmed mother's milk will be given to the skimmed mother's milk group. The fortifier is a standard fortifier we use in our population
  Arms: Skimmed mother's milk
Other: Specialized Formula — Infants will receive our standard of care - specialized formula
  Arms: Specialized Formula

SUMMARY:
The purpose of this study is to determine if the use of fortified skimmed mother's milk is a safe alternative to specialized formula in the treatment of chylothorax following cardiothoracic surgery.

DETAILED DESCRIPTION:
A chylothorax is a collection of fluid around the lungs that can occur after cardiac surgery. The fluid contains chyle, a milky fluid consisting of fat droplets. The standard treatment is to feed an infant with a specialized low fat formula for up to 6 weeks until the chest has time to heal. This formula is generally not well tolerated and mother's of our patients have expressed a desire to continue using breast milk. A few case reports have been published, but there have not been any studies to date looking at this. Data will be collected to include information about nutrition, weight gain, teaching needs, surgical, hospital, and discharge information.

ELIGIBILITY:
Inclusion Criteria:

* Infant birth to 12 months of age
* Undergo cardiothoracic surgery
* Develop a chylous effusion
* Be a breastfed or formula fed infant

Exclusion Criteria:

* Infant over 12 months of age
* Infant in state custody (foster care)
* Infant with milk protein allergy
* Infant born with congenital chylothorax
* Infant who develops chylothorax from other surgeries (non-cardiac

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the time to resolution of chylothorax of infants receiving skimmed mother's milk versus specialized formula. | up to 2 months from enrollment
  Fluid around the lungs is assessed by chest radiographs (x-rays) as per our usual standard of care. Cloudy fluid will be sent for analysis (chylomicrons, cell count, lymphocytes, and triglycerides) to confirm the diagnosis. The date of diagnosis, the date of chest tube removal, and the date of resolution of effusion by chest xrays

SECONDARY OUTCOMES:
To evaluate the recurrence rate of chylous effusion in infants receiving skimmed mother's milk versus specialized formula. | up to 4 months after hospital discharge
  All patients receive a standard chest x-ray prior to discharge from the hospital and again in two weeks at their follow up appointment. If symptoms of respiratory difficulty occur prior to or following this time, additional chest x-rays may be obtained based on exam findings and clinical judgment. The date of recurrence of effusion will be recorded as will the date of chest tube insertion if required.
To evaluate the technique of skimming and fortifying breast milk | the first 30 days after enrollment
  The skimming technique will be taught to participating mothers and nurses caring for their infants. A sample of the skim milk will be analyzed by a creamatocrit for fat and caloric content.
To compare feeding tolerance, growth, and nutrition in infants who receive fortified skimmed mother's milk versus specialized formula | 2 months
  Feeding symptoms observed by clinical staff and parents will be recorded. Parents will complete a questionnaire and score symptoms based on severity. Infants will be monitored as per our usual standard of care with weights, length measurements, and monitoring intake to ensure adequate growth

CONTACTS AND LOCATIONS:
Overall Officials: Cindi Farnstrom, MN, CPNP, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University - Doernbecher Children's Hospital, Portland, Oregon, United States

REFERENCES:
- [Background] Le Coultre C, Oberhansli I, Mossaz A, Bugmann P, Faidutti B, Belli DC. Postoperative chylothorax in children: differences between vascular and traumatic origin. J Pediatr Surg. 1991 May;26(5):519-23. doi: 10.1016/0022-3468(91)90696-q. PMID 2061800
- [Background] Milonakis M, Chatzis AC, Giannopoulos NM, Contrafouris C, Bobos D, Kirvassilis GV, Sarris GE. Etiology and management of chylothorax following pediatric heart surgery. J Card Surg. 2009 Jul-Aug;24(4):369-73. doi: 10.1111/j.1540-8191.2008.00781.x. PMID 19583606
- [Background] Chan EH, Russell JL, Williams WG, Van Arsdell GS, Coles JG, McCrindle BW. Postoperative chylothorax after cardiothoracic surgery in children. Ann Thorac Surg. 2005 Nov;80(5):1864-70. doi: 10.1016/j.athoracsur.2005.04.048. PMID 16242470
- [Background] Beghetti M, La Scala G, Belli D, Bugmann P, Kalangos A, Le Coultre C. Etiology and management of pediatric chylothorax. J Pediatr. 2000 May;136(5):653-8. doi: 10.1067/mpd.2000.104287. PMID 10802499
- [Background] Bond SJ, Guzzetta PC, Snyder ML, Randolph JG. Management of pediatric postoperative chylothorax. Ann Thorac Surg. 1993 Sep;56(3):469-72; discussion 472-3. doi: 10.1016/0003-4975(93)90881-h. PMID 8379718
- [Background] Suddaby EC, Schiller S. Management of chylothorax in children. Pediatr Nurs. 2004 Jul-Aug;30(4):290-5. PMID 15511045
- [Background] Allen EM, van Heeckeren DW, Spector ML, Blumer JL. Management of nutritional and infectious complications of postoperative chylothorax in children. J Pediatr Surg. 1991 Oct;26(10):1169-74. doi: 10.1016/0022-3468(91)90325-n. PMID 1779326
- [Background] Lessen R. Use of skim breast milk for an infant with chylothorax. ICAN: Infant, Child, & Adolescent Nutrition. 2009; 1(6):303-310.
- [Background] Chan GM, Lechtenberg E. The use of fat-free human milk in infants with chylous pleural effusion. J Perinatol. 2007 Jul;27(7):434-6. doi: 10.1038/sj.jp.7211768. Epub 2007 Jun 7. PMID 17554391
- [Background] Staats BA, Ellefson RD, Budahn LL, Dines DE, Prakash UB, Offord K. The lipoprotein profile of chylous and nonchylous pleural effusions. Mayo Clin Proc. 1980 Nov;55(11):700-4. PMID 7442324
- [Background] Cormack BE, Wilson NJ, Finucane K, West TM. Use of Monogen for pediatric postoperative chylothorax. Ann Thorac Surg. 2004 Jan;77(1):301-5. doi: 10.1016/s0003-4975(03)01189-5. PMID 14726083
- [Background] Orange JS, Geha RS, Bonilla FA. Acute chylothorax in children: selective retention of memory T cells and natural killer cells. J Pediatr. 2003 Aug;143(2):243-9. doi: 10.1067/S0022-3476(03)00305-6. PMID 12970641
- [Background] Sheeran T, Marvin RS, Pianta RC. Mothers' resolution of their child's diagnosis and self-reported measures of parenting stress, marital relations, and social support. J Pediatr Psychol. 1997 Apr;22(2):197-212. doi: 10.1093/jpepsy/22.2.197. PMID 9114643
- [Background] Wang CD, Chu PS, Mellen BG, Shenai JP. Creamatocrit and the nutrient composition of human milk. J Perinatol. 1999 Jul-Aug;19(5):343-6. doi: 10.1038/sj.jp.7200204. PMID 10685254
- [Background] Chatterjee R, Chatterjee S, Datta T, Roy B, Marimuthu P. Longitudinal study of human milk creamatocrit and weight gain in exclusively breastfed infants. Indian Pediatr. 1997 Oct;34(10):901-4. PMID 9567552
- [Background] Lucas A, Gibbs JA, Lyster RL, Baum JD. Creamatocrit: simple clinical technique for estimating fat concentration and energy value of human milk. Br Med J. 1978 Apr 22;1(6119):1018-20. doi: 10.1136/bmj.1.6119.1018. PMID 638579
- [Background] Buttiker V, Fanconi S, Burger R. Chylothorax in children: guidelines for diagnosis and management. Chest. 1999 Sep;116(3):682-7. doi: 10.1378/chest.116.3.682. PMID 10492271
- [Background] Lewis CC, Scott DE, Pantell RH, Wolf MH. Parent satisfaction with children's medical care. Development, field test, and validation of a questionnaire. Med Care. 1986 Mar;24(3):209-15. doi: 10.1097/00005650-198603000-00003. PMID 3951263
- [Background] Berseth CL, Mitmesser SH, Ziegler EE, Marunycz JD, Vanderhoof J. Tolerance of a standard intact protein formula versus a partially hydrolyzed formula in healthy, term infants. Nutr J. 2009 Jun 19;8:27. doi: 10.1186/1475-2891-8-27. PMID 19545360